CLINICAL TRIAL: NCT02674841
Title: Efficacy of Live Feedback to Increase Objectively Monitored Adherence to Prescribed, Home-based, Exercise Therapy-dosage in 15 to 19 Year Old Adolescents With Patellofemoral Pain. A Randomized Controlled Superiority Trial
Brief Title: Live Feedback to Increase Adherence in Adolescents With Patellofemoral Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Michael Skovdal Rathleff, Post.doc., Aalborg University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N-20150070
Record Dates: First submitted 2016-02-01; First posted 2016-02-05 (Estimated); Last update posted 2016-11-17 (Estimated); Status verified 2016-11

CONDITIONS: Patellofemoral Pain Syndrome; Musculoskeletal Disorders; Joint Diseases
Keywords: Adolescent; Physical therapy modalities; Exercise intervention; Auditive feedback; Visual feedback
MeSH Terms: conditions — Patellofemoral Pain Syndrome; Musculoskeletal Diseases; Joint Diseases | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Feedback group (Experimental): Receives live feedback on TUT and pulling force during exercises.
  Interventions: Other: Feedback on TUT; Other: Exercise
- Control group (Active Comparator): Receives no feedback on TUT but on pulling force during exercises.
  Interventions: Other: No feedback on TUT; Other: Exercise

INTERVENTIONS:
Other: Feedback on TUT — Access to live visual and auditory feedback on TUT and pulling force from an application on an iPad.
  Arms: Feedback group
Other: No feedback on TUT — Access only to live visual feedback on pulling force from an application on an iPad.
  Arms: Control group
Other: Exercise — 3 exercises (knee extension, hip abduction and hip extension) using an elastic band with 3 sets of 10 repetitions at 10-12 RM 3 times a week for 6 weeks.

SUMMARY:
This study investigates if live feedback during home-based exercises will improve the ability to perform the exercises with the prescribed time under tension (TUT) per repetition compared with no feedback among adolescents with patellofemoral pain. The hypothesis is that adolescents who receive live feedback from BandCizer™ will have a mean TUT that is significantly closer to the prescribed TUT compared to the group not receiving feedback during the course of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* 15 to 19 years of age
* Anterior knee pain of non-traumatic origin which is provoked by at least two of the following activities: prolonged sitting with bended knees or kneeling, squatting, running, jumping or ascending or descending stairs
* Tenderness on palpation of the peripatellar borders
* Pain of more than 6 weeks duration
* Worst pain during the previous week ≥ 30 mm on a 100 mm VAS

Exclusion Criteria:

* Concomitant pain from other structures in the knee (e.g. ligament, tendon or cartilage), the hip or the lumbar spine
* Previous knee surgery
* Patellofemoral instability

Ages: 15 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2016-02; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Mean deviation from the prescribed TUT per repetition in seconds during the course of the intervention | From 0-6 weeks
  The mean deviation is calculated as the difference between actual TUT and prescribed TUT (8 seconds). E.g. if the actual TUT is 6.5 seconds, the deviation is 1.5 seconds

SECONDARY OUTCOMES:
The total number of repetitions performed | From 0-6 weeks
Pulling force exerted per repetition measured in kilos | From 0-6 weeks
  This will be expressed as the maximum pulling force during each repetition
Isometric strength | At baseline and at the 6 week follow up
  Presented as Nm/kg in x, y and z direction
Pain measured on a 100 mm VAS | From 0-6 weeks
  Is entered into the app by the adolescent before and after each exercise
Kujala Patellofemoral Scale-score | At baseline and at the 6 week follow up
  Gives a score on patellofemoral pain ranging from 0 to 100 with 0 as complete disability and 100 as fully functional
Global rating of change | At the 6 week follow up
  Self-reported recovery on a 7-point Likert scale ranging from "much improved" to "much worse"
Summary of resistance | From 0-6 weeks
  Total pulling force exerted during the course of the intervention measured in kilos

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Rathleff, Ph.d., Principal Investigator — Aalborg University
Locations (1):
- Aalborg Universitetshospital, Aalborg, The North Denmark Region, Denmark

IPD SHARING:
Plan to Share IPD: Yes
No later than 1 year after the final follow-up, a completely anonymised data set to an appropriate data archive for sharing purposes will be delivered.

REFERENCES:
- [Derived] Riel H, Matthews M, Vicenzino B, Bandholm T, Thorborg K, Rathleff MS. Efficacy of live feedback to improve objectively monitored compliance to prescribed, home-based, exercise therapy-dosage in 15 to 19 year old adolescents with patellofemoral pain- a study protocol of a randomized controlled superiority trial (The XRCISE-AS-INSTRUcted-1 trial). BMC Musculoskelet Disord. 2016 Jun 2;17:242. doi: 10.1186/s12891-016-1103-y. PMID 27250984